CLINICAL TRIAL: NCT02340130
Title: A Multicentre, Open Label, Phase IIb Clinical Trial to Evaluate Safety, Tolerability and Efficacy of the Depigmented Modified Allergen Extract of Two Mites Mixes at 200 DPP/ml (DP/MG/14-1 Dermatophagoides Pteronyssinus / Lepidoglyphus Destructor and DP/MG/14-2 Dermatophagoides Pteronyssinus /Blomia Tropicalis) in Subjects With Allergic Rhinitis or Rhinoconjunctivitis, With Controlled Allergic Asthma
Brief Title: Safety, Tolerability and Efficacy of the Depigmented Modified Allergen Extract of Two Mites in Subjects With Allergic Rhinitis or Rhinoconjunctivitis, With Controlled Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301-PG-PSC-203
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis; Rhinoconjunctivitis; Asthma
MeSH Terms: conditions — Rhinitis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DP/MG/14-1 (Experimental): DP/MG/14-1: Depigmented modified allergen extract of D. pteronyssinus 50% / Depigmented, glutaraldehyde-polymerised B. tropicalis 50% (200DPP/mL) The administration regimen will consist of a rush build-up régimen and a follow up period
  Interventions: Biological: DP/MG/14-1
- DP/MG/14-2 (Experimental): DP/MG/14-2: Depigmented modified allergen extract of D. pteronyssinus 50% / Depigmented, glutaraldehyde-polymerised L.destructor 50% (200DPP/mL) The administration regimen will consist of a rush build-up régimen and a follow up period
  Interventions: Biological: DP/MG/14-2

INTERVENTIONS:
Biological: DP/MG/14-1 — The administration regimen will consist of a rush build-up régimen and a follow up period
  Arms: DP/MG/14-1
Biological: DP/MG/14-2 — The administration regimen will consist of a rush build-up régimen and a follow up period
  Arms: DP/MG/14-2

SUMMARY:
This is an open-label, non-controlled, non-randomised, prospective safety study in patients with rhinitis or allergic rhinoconjunctivitis, with controlled asthma, and clinically relevant sensitisation to dust mites from the Pyroglyphidae and Glycyphagidae families.

DETAILED DESCRIPTION:
The objective is to evaluate the safety and tolerability of the administration of two allergen extracts of dust mite mixtures at 200 DPP/ml (DP/MG/14-1 Dermatophagoides pteronyssinus / Blomia tropicalis and DP/MG/14-2 Dermatophagoides pteronyssinus / Lepidoglyphus destructor) using a rush build-up phase in patients with allergic rhinitis or rhinoconjunctivitis, with controlled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided appropriately signed and dated written informed consent.
2. Men and women aged 18 years and 70 years of age at Visit 1.
3. Has an FEV1 value 80% of predicted normal value at Visit 1.
4. Individuals suffering from perennial allergic rhinitis or rhinoconjunctivitis moderate-severe for at least the preceding year, with controlled asthma, caused by double sensitization against Dermatophagoides pteronyssinus (DPT) and Lepidoglyphus destructor or Dermatophagoides pteronyssinus and Blomia tropicalis.
5. Patients sensitized to co-allergens such as tree pollen, grasses or weeds, fungi or animal epithelials cannot participate in the study if they are symptomatic.
6. If a female is of non-childbearing potential, the subject must be postmenopausal for at least 1 year or surgically sterile.
7. If a female is of childbearing potential, the subject must be non-lactating and non-pregnant and must correctly use an effective method of contraception during the study.

Exclusion Criteria:

1. Any contraindication for treatment with allergen specific immunotherapy.
2. Subjects with a previous history of anaphylaxis.
3. Patients with hospital admission due to asthma exacerbations within 1 year prior to V1.
4. Has uncontrolled asthma, according to Global Initiative for Asthma Guidelines (GINA 2010).
5. Acute or chronic infectious conjunctivitis.
6. Has acute or chronic inflammatory or infectious airways disease.
7. Has chronic structural diseases of the affected organ (e.g. eye, nose, lung).
8. History or presence of confirmed or potential diseases of the immune system including autoimmune diseases and immune deficiencies of actual clinical relevance.
9. Has any disease that prohibits the use of adrenaline (e.g., hyperthyroidism).
10. Has a severe uncontrolled disease that could increase the risk to the subjects while participating in the study, including but not limited to, the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases or haematological disord

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Subjects (%) suffering from immediate or delayed systemic grade 2 reactions | Safety: local and systemic adverse reactions (EAACI classification) within 24 and 48 hours after the treatment.
  Subjects (%) suffering from immediate or delayed systemic grade 2 reactions, according to EACCI 2006 classification, along the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Sanchez, Study Chair — Laboratorios Leti, S.L.U
Locations (3):
- Spain (3):
  - Hospital de Conxo, Santiago de Compostela, A Coruña
  - Hosp Ntra Sra de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Lucus-Augusti, Lugo